CLINICAL TRIAL: NCT06162650
Title: A Phase II Study of Total Neoadjuvant Therapy in Rectal Cancer
Brief Title: Total Neoadjuvant Therapy in Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Min Yeh, MD, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-112-042
Record Dates: First submitted 2023-11-27; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Consolidation Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): The total neoadjuvant therapy with the short-course radiotherapy (5×5 Gy over a maximum of 8 days) followed by chemotherapy with mFOLFOX6 for 9 cycles will be administered.
  Interventions: Radiation: Short-course radiotherapy; Drug: mFOLFOX6

INTERVENTIONS:
Radiation: Short-course radiotherapy — Short-course radiotherapy, 5×5 Gy.
  Other Names: RT
Drug: mFOLFOX6 — Oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, infusinal 5-fluorouracil 2400 mg/m2 every 2 weeks, for 9 cycles
  Other Names: Consolidation chemotherapy

SUMMARY:
In this phase 2 study, the efficacy of total neoadjuvant therapy in Taiwanese patients with rectal cancer will be investigated. Patients with stage II or III middle/low rectal cancer will be prospective enrolled. The total neoadjuvant therapy with the short-course radiotherapy (5×5 Gy over a maximum of 8 days) followed by chemotherapy with mFOLFOX6 for 9 cycles will be administered. The primary endpoint is the complete response (CR) rate which will take into account the patients with clinical and pathological complete response.

DETAILED DESCRIPTION:
This is a single center, single-arm, open-label, phase II study to investigate the efficacy and toxicities of total neoadjuvant therapy in patients with middle or lower rectal cancer. This study is planned to start after the approval by IRB, enroll patients for 2 years, and follow the clinical outcome for another 5 years. It will be conducted at National Cheng Kung University Hospital. Forty-two subjects will be enrolled. Patients who have newly diagnosed stage II or III, middle or low rectal adenocarcinoma will be recruited to receive the TNT treatment. The TNT includes the short-course radiotherapy (5×5 Gy over a maximum of 8 days)) followed by chemotherapy with the regimen of mFOLFOX6 for total 9 cycles

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the rectum;
* Tumors located at mid or low rectum (distal extension less than 10 cm from the anal verge);
* Clinical stage II or III (T3/4 and/or N+; no distant metastasis);
* No prior chemotherapy, radiotherapy or surgery for rectal cancer;
* Age ≥20;
* ECOG 0-1;
* Adequate organ function, including followings:

ANC ≥1,500/μL; Hb ≥8.0 gm/dL; Platelet 100,000/mm3; Total bilirubin ≤1.5x upper normal limit; AST ≤3x upper normal limit; ALT ≤3x upper normal limit; Creatinine ≤1.5x upper normal limit;

* Ability to understand and the willingness to sing a written informed consent.

Exclusion criteria

* Recurrent rectal cancer;
* Patients who have concomitant malignancies, except for adequately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix. Subjects who have prior malignancies and have been disease-free for more than 5 years can be enrolled;
* Patients who have received prior pelvic radiotherapy;
* Patients with active infection requiring intravenous antibiotic treatment;
* Patients with a history of any arterial thrombotic event within the past 6 months, including unstable angina, myocardial infarction (MI) or cerebrovascular accident (CVA), New York Hear Association (NYHA) grade II or greater congestive heart failure, or uncontrolled cardiac arrhythmia;
* Patients with any other concurrent medical or psychiatric condition or disease which, in the investigator's judgement, would make them inappropriate candidates for entry into this study;
* Women who are pregnant or breastfeeding. Women of childbearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period;
* Patients receiving other anticancer or experimental therapy;
* Known DPD deficiency or hypersensitivity to oxaliplatin;
* Any contraindications to MRI.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-11-16 (Estimated); Study Completion 2030-11-16 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | The response will be assessed at the period of 2 to 4 weeks after the completion of total neoadjuvant chemotherapy
  The percentage of patients who achieve a complete response

SECONDARY OUTCOMES:
R0 resection rate | The R0 resection rate will be assessed at the period of 2 to 4 weeks after completion of the total neoadjuvant chemotherapy
  The percentage of patients who receive the surgery of total neoadjuvant therapy and achieve R0 resection
Response rate | The response will be assessed at the period of 2 to 4 weeks after the completion of total neoadjuvant chemotherapy
  The percentage of patients who achieve a complete response or partial response
Loco-regional failure rate | The loco-regional failure will be assessed from the date of surgical resection until the first documented local recurrence, up to 84 months
  The percentage of patients who develop local recurrence after surgery
Rate of distant metastasis | The distant metastasis will be assessed from the date of beginning short-course RT until the first documented distant metastasis, up to 84 months
  The percentage of patients who develop distant metastasis
Safety profiles | The safety profile will be assessed from the beginning of the short-course RT to the end of last cycle of FOLFOX chemotherapy, up to 24 weeks
  The occurrence and severity of adverse events which develop during the treatment of total neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Min Yeh, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan